CLINICAL TRIAL: NCT07002060
Title: A Phase 3 Randomized, Modified Double-blind, Active-controlled Study to Assess the Safety of vYF, Yellow Fever Vaccine, in Adults Aged 18 Years up to 60 Years
Brief Title: Phase 3 Randomized, Modified Double-blind, Active-controlled Safety Study on vYF in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYF00019
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Yellow Fever Immunization
Keywords: Yellow fever
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Sponsor study staff, investigators and study staff, will remain blinded during the study conduct, except dedicated study staff preparing/administering the study interventions and who are not involved in the safety evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vYF vaccine (Experimental): A single dose on Day 01
  Interventions: Biological: Yellow fever vaccine (live)
- YF-VAX vaccine (Active Comparator): A single dose on Day 01
  Interventions: Biological: YF vaccine (live)

INTERVENTIONS:
Biological: Yellow fever vaccine (live) — Powder and solvent for solution for injection Subcutaneous
  Other Names: vYF vaccine
  Arms: vYF vaccine
Biological: YF vaccine (live) — Powder and diluent for suspension for injection Subcutaneous
  Other Names: YF-VAX vaccine; YF-VAX
  Arms: YF-VAX vaccine

SUMMARY:
The purpose of this study is to assess the safety of vYF (investigational vaccine) compared to the safety of YF-VAX (YF licensed vaccine) in adults aged 18 years up to 60 years.

Study details include:

* The study duration will be up to approximately 6 months.
* One single dose of the study intervention (vYF or YF-VAX) will be administered subcutaneously at the 1st visit.
* The visit(V) frequency will be Day(D) 01 (V01) and D29 (V02). Two telephone calls will be planned at D15 and Month(M)6.

Number of Participants:

A total of 640 participants are expected to be included in the study in a 3:1 ratio (vYF: YF-VAX):

Group 1: vYF; N=480 Group 2: YF-VAX; N=160

Study Arms and Duration:

Randomized, active control (YF-VAX). 6 months duration per participants. Eligible participants will be randomized in a 3:1 ratio to receive, subcutaneously, a single dose of vYF or YF-VAX vaccines on D01.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 years to 60 years on the day of inclusion
* Participants who are healthy as determined by medical evaluation including medical history and physical examination
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, or surgically sterile.

OR

-Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) before any dose of study intervention on D01 and will be repeated on D29 to confirm the participant is still not pregnant within the 28 days of vaccine administration
* Able to attend all scheduled visits and to comply with all study procedures Informed consent
* Informed consent form has been signed and dated

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known history of laboratory evidence of HIV infection
* Known history of hepatitis B or hepatitis C seropositivity
* Known history of flavivirus (FV) infection
* Known systemic hypersensitivity to any of the study intervention components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances
* Personal or family history of thymic pathology (thymoma, thymectomy, or myasthenia)
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion , including malignancy, such as leukemia or lymphoma
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38°C [or ≥ 100.4°F]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination (prior to Visit 2 on D29), except for influenza vaccination, which may be received at least 2 weeks before study vaccine. This exception includes pandemic influenza vaccines including monovalent pandemic influenza vaccines.
* Previous vaccination against a FV disease at any time including yellow fever (YF) with an investigational or marketed vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 6 months
* Administration of any anti-viral within 2 months preceding the vaccination and up to the 6 weeks following the vaccination
* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the course of the study in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Planned travel in a YF endemic country within 6 months of investigational vaccine administration

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 640 (Actual)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events are any unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site reactions | Up to 7 days after vaccination
  Solicited injection site reactions include injection site pain, erythema and swelling
Number of participants with solicited systemic reactions | Up to 14 days after vaccination
  Solicited systemic reactions include fever, headache, malaise and myalgia
Number of participants with unsolicited adverse events (AEs) | Up to 28 days after vaccination
  Unsolicited (spontaneously reported) AEs, not fulfilling criteria for solicited adverse reactions
Number of participants with medical attended adverse events (MAAEs) | Up to 28 days after vaccination
  MAAEs
Number of participants with adverse events of special interest (AESIs) | Up to 6 months after vaccination
  AESIs
Number of participants with serious adverse events (SAEs) | Up to 6 months after vaccination
  SAEs

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - The Hope Clinic of Emory University- Site Number : 8400006, Decatur, Georgia
  - Velocity Clinical Research-New Orleans- Site Number : 8400004, New Orleans, Louisiana
  - Johns Hopkins Bloomberg School of Public Health- Site Number : 8400009, Baltimore, Maryland
  - Saint Louis University Center for Vaccine Development- Site Number : 8400001, St Louis, Missouri
  - Rochester Clinical Research- Site Number : 8400005, Rochester, New York
  - Velocity Clinical Research - Providence- Site Number : 8400003, East Greenwich, Rhode Island
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VYF00019 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26722&tenant=MT_SNY_9011